CLINICAL TRIAL: NCT07288762
Title: Gonadal Function in Boys With Transfusion Depandant Beta Thalassemia
Brief Title: Gonadal Function in Thalassemic Patient
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hager Saadeldin Mohamed, pediatric resident, Sohag University
Other Study IDs: Soh-Med-25-9-18MS
Record Dates: First submitted 2025-11-22; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Thalassemia Majors (Beta-Thalassemia Major)
Keywords: INSL3 or inhibin B hormone in transfusion depandant beta thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1 transfusion depandant beta thalassemia: transfusion depandant beta thalassemia 10 - 18 years old age gonadal function assesment
  Interventions: Diagnostic Test: serum inhibin B serum INSL3 serum AMH

INTERVENTIONS:
Diagnostic Test: serum inhibin B serum INSL3 serum AMH — transfusion depandant beta thalassemia with measure gonadal function serum INSL3 serum inhibin B serum AMH

SUMMARY:
Patient with transfusion depandant beta thalassemia with accumulation of iron in their body affect pituitary gland and gonades lead to impaired their functions .

DETAILED DESCRIPTION:
detection of any abnormalities in pituitary gland hormones ( FSH , LH , serum prolactin ) gonadal hormones ( serum testesterone , antimullerian hormone , INSL3 , inhibin B hormone )

ELIGIBILITY:
Inclusion Criteria:

* transfusion depandant beta thalassemia
* age 10 to 18 year old age

Exclusion Criteria:

* age below 10 year old age or above 18 year old age
* associated with another disease

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: transfusion depandant beta thalassemia male patients age 10 - 18 year old age
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
gonadal function in transfusion depandant beta thalassemia | through study completion, an average of 1 year
  gonadal function assessment by Inhibin B hormone, INSL3 , serum testesterone that analysed in patient with age 10 - 18 year old for early detection of any abnormality

CONTACTS AND LOCATIONS:
Overall Officials: hager Saadeldin, resident, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided